CLINICAL TRIAL: NCT03980223
Title: Evaluation of Doxycycline Post-exposure Prophylaxis to Reduce Sexually Transmitted Infections in PrEP Users and HIV-infected Men Who Have Sex With Men
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Washington (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Mayne Pharma International Pty Ltd (Industry); San Francisco Department of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DoxyPEP; R01AI143439 (NIH)
Record Dates: First submitted 2019-06-06; First posted 2019-06-10 (Actual); Results first posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-06

CONDITIONS: Gonorrhea; Chlamydia; Syphilis
Keywords: HIV; Post-Exposure Prophylaxis; Men who have sex with men (MSM); Doxycycline; HIV Pre-Exposure Prophylaxis; Sexually transmitted infection
MeSH Terms: conditions — Gonorrhea; Chlamydia Infections; Syphilis; Homosexuality; Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: Open-label randomized clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Doxy PEP (Experimental): Doxycycline 200mg in addition to standard of care STI testing and treatment
  Interventions: Drug: Doxycycline Hyclate Delayed-Release 200 mg
- Control (No Intervention): The control arm will consist of standard of care STI testing and treatment

INTERVENTIONS:
Drug: Doxycycline Hyclate Delayed-Release 200 mg — 200 mg of doxycycline taken by mouth after condomless sexual contact as post exposure prophylaxis (PEP)
  Arms: Doxy PEP

SUMMARY:
The purpose of this study is to understand if taking an antibiotic called doxycycline by mouth as soon as possible after sexual contact without a condom can reduce the risk of sexually transmitted infections (STIs), including gonorrhea, chlamydia and syphilis. The study will also look at the safety of doxycycline PEP and the impact that PEP may have on the bacteria that cause STIs as well as on bacteria that normally live on the body. While doxycycline is approved by the Food and Drug Administration (FDA), taking doxycycline immediately after sexual contact to prevent infection is investigational and is not approved by the FDA for this use. Participants will take part in the study for 1 year.

DETAILED DESCRIPTION:
The overarching goal is to assess the effectiveness of doxycycline PEP on incidence of STIs and tetracycline resistance among STIs and commensal bacteria to inform public health policy. Participants will be randomized 2:1, with a greater number receiving doxycycline PEP compared with the standard of care control, to maximize data on safety, tolerability, adherence coverage of sexual acts, and resistance data in participants randomized to doxycycline PEP, without negatively impacting power to measure effectiveness. Participants will be counseled about the preliminary effectiveness data from IPERGAY, and the potential for antimicrobial resistance (AMR) in STIs or other bacteria. Possibility of unreported doxycycline us in the control arm (contamination) will be monitored through retrospective batch testing of doxycycline metabolites in hair, to detect doxycycline use in the prior 3 months. 53

Eligible participants randomized 2:1 to receive PEP will receive open-label doxycycline 200 mg to be taken ideally within 24 hours but no later than 72 hours after condomless sexual contact (oral or anal). 200 mg of doxycycline will be taken at most once per 24 hour period regardless of the number of sexual acts occurring during this time period. Sexual activity will be recorded for both arms of the study (doxycycline PEP and control condition) by the participant using a smartphone application that will be adapted for study use; this will enable comparable assessment of risk in the two arms. PEP pill-taking will also be measured by the app to enable assessment of coverage of sex acts by PEP. Sexual activity and adherence will also be assessed in person at quarterly visits. STI testing will be conducted quarterly from three anatomic sites (pharyngeal, rectal and urinary) and blood for syphilis testing. Participants with a positive STI test will return for STI treatment and for swabs of the affected site for resistance testing; culture based for gonorrhea (GC) and molecular methods for CT and syphilis. Those with a serologic test that indicates a new syphilis infection will have swabs of any current active lesion as well as mucosal swabs from the oropharynx. Nares and oropharyngeal swabs will be obtained at baseline, 6 and 12 months to evaluate tetracycline resistance in S. aureus among carriers and in commensal Neisseria species.

Stool samples from 100 participants on the doxycycline PEP arm - 50 MSM living with HIV and 50 HIV uninfected MSM on pre-exposure prophylaxis (PrEP) - will be collected at baseline, 6 and 12 months to evaluate effects of intermittent doxycycline on the gut resistome, using 16s ribosomal RNA amplification to study tetracycline resistance genes. Rectal swabs will be collected and archived in all participants at baseline, 6, and 12 months for future studies of the impact of doxycycline PEP on the enteric microbiome and resistome.

Study population: This study will enroll 390 HIV-infected participants and 390 persons taking PrEP, for a total sample size of 780. An approximately equal number of participants in each of these cohorts (and in each study arm) will be enrolled in San Francisco and Seattle.

Current or planned initiation of PrEP use is an eligibility criterion for enrollment, because this population of MSM has high rates of STIs and are typically seen quarterly for PrEP visits. However, participants may opt to stop PrEP use at any time during the study without affecting their involvement in the study. Any HIV-uninfected participants who subsequently seroconvert will be managed clinically by the study site according to local practice (appropriate counseling, clinical evaluation and immediate linkage to clinical and psychosocial services). These participants will also be retained in the study unless they choose to discontinue study participation.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent
* Age ≥ 18 years
* Male sex at birth
* Previously HIV-diagnosed OR HIV-seronegative at the time of last test within the past month and a current prescription for PrEP (both daily or event-driven permitted) or plan to start PrEP within 30 days after the enrollment visit
* Condomless anal or oral sexual contact with ≥ 1 male sex-at-birth partners in the past 12 months
* Diagnosed with GC, CT or early syphilis (primary, secondary or early latent) in the past 12 months. Note: self report of STI is acceptable if documentation not available. If the participant reports an incident STI in the past year at the same clinic where the participant will be enrolled, this diagnosis should be confirmed by chart review prior to enrollment. If the diagnosis from this clinic cannot be confirmed, the participant should not be enrolled. If the STI was reported at a clinical site that is not the study site, and records cannot be obtained, self-report will suffice.

Note: Syphilis diagnosis within the last year refers to primary syphilis, secondary syphilis, and documented early latent syphilis (< 1 year since last syphilis diagnosis or negative test). Known late latent syphilis or latent syphilis of unknown duration would not qualify. Positive syphilis titers which represent serofast status and not active disease do not qualify as a syphilis diagnosis. Clinician judgement regarding qualifying syphilis diagnosis should be sought when the diagnosis of syphilis in the past year is not clear or if there is a question about serofast status vs. active infection.

Exclusion Criteria:

* Allergy to tetracycline class
* Current medications which may impact doxycycline metabolism or that are contraindicated with doxycycline, as per the prescribing information. These include systemic retinoids, barbiturates, carbamazepine, and phenytoin.
* Current use of warfarin, as intermittent doxycycling use can lead to an unpredictable impact on INR
* Anticipated use of doxycycline during the coming 12 months for non-STI prevention (e.g., acne treatment).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 641 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Luetkemeyer, MD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - San Francisco City Clinic / San Francisco Department of Public Health, San Francisco, California
  - University of California, San Francisco / Zuckerberg San Francisco General Hospital/UCSF, San Francisco, California
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers outside of the study team

REFERENCES:
- [Background] Molina JM, Charreau I, Chidiac C, Pialoux G, Cua E, Delaugerre C, Capitant C, Rojas-Castro D, Fonsart J, Bercot B, Bebear C, Cotte L, Robineau O, Raffi F, Charbonneau P, Aslan A, Chas J, Niedbalski L, Spire B, Sagaon-Teyssier L, Carette D, Mestre SL, Dore V, Meyer L; ANRS IPERGAY Study Group. Post-exposure prophylaxis with doxycycline to prevent sexually transmitted infections in men who have sex with men: an open-label randomised substudy of the ANRS IPERGAY trial. Lancet Infect Dis. 2018 Mar;18(3):308-317. doi: 10.1016/S1473-3099(17)30725-9. Epub 2017 Dec 8. PMID 29229440
- [Background] The Lancet Hiv. U=U taking off in 2017. Lancet HIV. 2017 Nov;4(11):e475. doi: 10.1016/S2352-3018(17)30183-2. No abstract available. PMID 29096785
- [Background] Harrison WO, Hooper RR, Wiesner PJ, Campbell AF, Karney WW, Reynolds GH, Jones OG, Holmes KK. A trial of minocycline given after exposure to prevent gonorrhea. N Engl J Med. 1979 May 10;300(19):1074-8. doi: 10.1056/NEJM197905103001903. PMID 107450
- [Background] Steen R, Chersich M, Gerbase A, Neilsen G, Wendland A, Ndowa F, Akl EA, Lo YR, de Vlas SJ. Periodic presumptive treatment of curable sexually transmitted infections among sex workers: a systematic review. AIDS. 2012 Feb 20;26(4):437-45. doi: 10.1097/QAD.0b013e32834ed991. PMID 22095197
- [Background] Bolan RK, Beymer MR, Weiss RE, Flynn RP, Leibowitz AA, Klausner JD. Doxycycline prophylaxis to reduce incident syphilis among HIV-infected men who have sex with men who continue to engage in high-risk sex: a randomized, controlled pilot study. Sex Transm Dis. 2015 Feb;42(2):98-103. doi: 10.1097/OLQ.0000000000000216. PMID 25585069
- [Background] Sloan B, Scheinfeld N. The use and safety of doxycycline hyclate and other second-generation tetracyclines. Expert Opin Drug Saf. 2008 Sep;7(5):571-7. doi: 10.1517/14740338.7.5.571. PMID 18759709
- [Background] Turner RB, Smith CB, Martello JL, Slain D. Role of doxycycline in Clostridium difficile infection acquisition. Ann Pharmacother. 2014 Jun;48(6):772-6. doi: 10.1177/1060028014528792. Epub 2014 Mar 28. PMID 24682682
- [Background] Nadelman RB, Nowakowski J, Fish D, Falco RC, Freeman K, McKenna D, Welch P, Marcus R, Aguero-Rosenfeld ME, Dennis DT, Wormser GP; Tick Bite Study Group. Prophylaxis with single-dose doxycycline for the prevention of Lyme disease after an Ixodes scapularis tick bite. N Engl J Med. 2001 Jul 12;345(2):79-84. doi: 10.1056/NEJM200107123450201. PMID 11450675
- [Background] Angelakis E, Armstrong N, Nappez C, Richez M, Chabriere E, Raoult D. Doxycycline assay hair samples for testing long-term compliance treatment. J Infect. 2015 Nov;71(5):511-7. doi: 10.1016/j.jinf.2015.08.003. Epub 2015 Aug 20. PMID 26299894
- [Derived] Luetkemeyer AF, Donnell D, Cohen SE, Dombrowski JC, Grabow C, Haser G, Brown C, Cannon C, Malinski C, Perkins R, Nasser M, Lopez C, Suchland RJ, Vittinghoff E, Buchbinder SP, Scott H, Charlebois ED, Havlir DV, Soge OO, Celum C. Doxycycline to prevent bacterial sexually transmitted infections in the USA: final results from the DoxyPEP multicentre, open-label, randomised controlled trial and open-label extension. Lancet Infect Dis. 2025 Aug;25(8):873-883. doi: 10.1016/S1473-3099(25)00085-4. Epub 2025 Mar 24. PMID 40147465
- [Derived] Chu VT, Glascock A, Donnell D, Grabow C, Brown CE, Ward R, Love C, Kalantar KL, Cohen SE, Cannon C, Woodworth MH, Kelley CF, Celum C, Luetkemeyer AF, Langelier CR. Impact of doxycycline post-exposure prophylaxis for sexually transmitted infections on the gut microbiome and antimicrobial resistome. Nat Med. 2025 Jan;31(1):207-217. doi: 10.1038/s41591-024-03274-2. Epub 2024 Oct 3. PMID 39363100
- [Derived] Fredericksen RJ, Perkins R, Brown CE, Cannon C, Lopez C, Cohee A, Dombrowski JC, Cohen S, Malinski C, Powell M, Luetkemeyer AF, Celum C, Christopoulos K. Doxycycline as Postsexual Exposure Prophylaxis: Use, Acceptability, and Associated Sexual Health Behaviors Among a Multi-Site Sample of Clinical Trial Participants. AIDS Patient Care STDS. 2024 Apr;38(4):155-167. doi: 10.1089/apc.2023.0289. PMID 38656217
- [Derived] Luetkemeyer AF, Donnell D, Dombrowski JC, Cohen S, Grabow C, Brown CE, Malinski C, Perkins R, Nasser M, Lopez C, Vittinghoff E, Buchbinder SP, Scott H, Charlebois ED, Havlir DV, Soge OO, Celum C; DoxyPEP Study Team. Postexposure Doxycycline to Prevent Bacterial Sexually Transmitted Infections. N Engl J Med. 2023 Apr 6;388(14):1296-1306. doi: 10.1056/NEJMoa2211934. PMID 37018493

RESULTS

PARTICIPANT FLOW:
Groups:
- PrEP Cohort: Doxy PEP: Doxycycline 200mg in addition to standard of care STI testing and treatment - HIV-negative participants on PrEP at time of enrollment or starting PrEP within 30 days of enrollment.
  Doxycycline Hyclate Delayed-Release 200 mg: 200 mg of doxycycline taken by mouth after condomless sexual contact as post exposure prophylaxis (PEP)
- PrEP Cohort: Control; PLWH: Control: The control arm will consist of standard of care STI testing and treatment - HIV-negative participants on PrEP at time of enrollment or starting PrEP within 30 days of enrollment.
- PLWH Cohort: Doxy PEP: Doxycycline 200mg in addition to standard of care STI testing and treatment - People living with HIV
  Doxycycline Hyclate Delayed-Release 200 mg: 200 mg of doxycycline taken by mouth after condomless sexual contact as post exposure prophylaxis (PEP)
Period: Overall Study
Arm/Group | PrEP Cohort: Doxy PEP | PrEP Cohort: Control | PLWH Cohort: Doxy PEP | PLWH: Control
Started | 292 | 140 | 141 | 68
Completed | 217 | 100 | 109 | 47
Not Completed | 75 | 40 | 32 | 21
Not completed — Lost to Follow-up | 3 | 7 | 10 | 8
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 2
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Not included because they had not yet reached month 3 visit at time of analysis | 72 | 33 | 20 | 11

BASELINE CHARACTERISTICS:
Population: Overall number of baseline participants does not include participants who had not yet reached their month 3 visit at the time of the analysis and those who were lost to FU after month 3.
Groups:
- PLWH Cohort: Control: The control arm will consist of standard of care STI testing and treatment - People living with HIV
- Total: Total of all reporting groups
Arm/Group | PrEP Cohort: Doxy PEP | PrEP Cohort: Control | PLWH Cohort: Doxy PEP | PLWH Cohort: Control | Total
Number analyzed (Participants) | 220 | 107 | 119 | 55 | 501
Age, Customized [Median (Inter-Quartile Range); unit: Years]
  Median age | 36 [31 to 42] | 36 [31 to 42] | 43 [36 to 54] | 42 [37 to 50] | 38 [32 to 47]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender identity: Man | 212 | 107 | 109 | 54 | 482
  Gender identity: Transgender woman or gender-diverse | 8 | 0 | 10 | 1 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 55 | 41 | 41 | 14 | 151
  Not Hispanic or Latino | 165 | 66 | 78 | 41 | 350
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Data not available for 19 participants.
  Participants
    Race: number analyzed (Participants) | 209 | 104 | 116 | 53 | 482
    Race: White | 144 | 66 | 74 | 37 | 321
    Race: Black | 9 | 5 | 15 | 7 | 36
    Race: Asian or Pacific Islander | 33 | 12 | 7 | 1 | 53
    Race: Multiple races or other | 23 | 21 | 20 | 8 | 72
Region of Enrollment [Number; unit: participants]
  United States | 220 | 107 | 119 | 55 | 501
Gender of sexual partners [Count of Participants; unit: Participants] — Population: Data not available for 1 participant.
  Participants
    number analyzed (Participants) | 220 | 107 | 118 | 55 | 500
    Men only | 191 | 90 | 105 | 48 | 434
    Multiple genders | 29 | 17 | 13 | 7 | 66
Annual income [Count of Participants; unit: Participants] — Population: Data not available for 2 participants.
  Participants
    number analyzed (Participants) | 219 | 106 | 119 | 55 | 499
    <$20,000 | 31 | 13 | 42 | 17 | 103
    $20,001-$50,000 | 64 | 39 | 40 | 22 | 165
    $50,001-$75,000 | 45 | 14 | 22 | 5 | 86
    >$75,000 | 79 | 40 | 15 | 11 | 145
STI in the past 12 months [Count of Participants; unit: Participants]
  Gonorrhea | 155 | 78 | 71 | 39 | 343
  Chlamydia | 144 | 63 | 58 | 27 | 292
  Syphillis | 32 | 16 | 35 | 17 | 100
Two or more STIs in the past 12 months [Count of Participants; unit: Participants] | 106 | 44 | 39 | 26 | 215
STI at baseline [Count of Participants; unit: Participants] — Population: Data was not available for participants as follows:
  * Gonorrhea: 5 participants
  * Chlamydia: 4 participants
  * Syphilis: 3 participants
  * Any STI: 7 participants
  Participants
    Gonorrhea: number analyzed (Participants) | 218 | 107 | 117 | 54 | 496
    Gonorrhea | 40 | 20 | 25 | 14 | 99
    Chlamydia: number analyzed (Participants) | 219 | 107 | 117 | 54 | 497
    Chlamydia | 31 | 11 | 11 | 8 | 61
    Syphilis: number analyzed (Participants) | 219 | 107 | 117 | 55 | 498
    Syphilis | 5 | 1 | 11 | 4 | 21
    Any STI at baseline: number analyzed (Participants) | 219 | 106 | 114 | 55 | 494
    Any STI at baseline | 65 | 27 | 34 | 20 | 146
Median number of sexual partners in past 3 months [Median (Inter-Quartile Range); unit: partners] | 8 [4 to 17] | 10 [5 to 16.5] | 7 [3 to 18.5] | 10.5 [3 to 20] | 9 [4 to 17]
Transactional sex during lifetime [Count of Participants; unit: Participants] — Population: Data not available for 10 participants
  Participants
    number analyzed (Participants) | 219 | 107 | 116 | 49 | 491
    (all) | 47 | 28 | 47 | 21 | 143
Substance use in the past 3 months [Count of Participants; unit: Participants] — Population: Data not available for 8 participants.
  Participants
    Stimulants: methamphetamine, cocaine, or crack: number analyzed (Participants) | 216 | 107 | 117 | 53 | 493
    Stimulants: methamphetamine, cocaine, or crack | 51 | 22 | 50 | 23 | 146
    Heroin or other opioids: number analyzed (Participants) | 216 | 107 | 117 | 53 | 493
    Heroin or other opioids | 2 | 1 | 9 | 2 | 14
    Ecstasy, GHB, or ketamine: number analyzed (Participants) | 216 | 107 | 117 | 53 | 493
    Ecstasy, GHB, or ketamine | 63 | 34 | 39 | 21 | 157
    Amyl nitrates, also known as poppers: number analyzed (Participants) | 216 | 107 | 117 | 53 | 493
    Amyl nitrates, also known as poppers | 93 | 47 | 56 | 28 | 224
    Marijuana: number analyzed (Participants) | 216 | 107 | 117 | 53 | 493
    Marijuana | 96 | 56 | 60 | 27 | 239
    Total with any substance use in past 3 months: number analyzed (Participants) | 216 | 107 | 117 | 53 | 493
    Total with any substance use in past 3 months | 112 | 66 | 77 | 38 | 293

OUTCOME MEASURES:

1. Primary Outcome: Number of Quarterly Visits In Which an STI Was Detected
Description: Number of quarterly visits with an STI event detected.
Time Frame: 1 year
Population: Primary efficacy analysis population excludes participants who did not attend any follow-up visits after baseline.
Measure: Number; unit: No. quarterly visits with STI event
Units Other Than Participants: Total number of quarterly visits
Arm/Group | PrEP Cohort: Doxy PEP | PrEP Cohort: Control | PLWH Cohort: Doxy PEP | PLWH: Control
Number analyzed (Participants) | 217 | 100 | 109 | 47
Number analyzed (Total number of quarterly visits) | 570 | 257 | 305 | 128
No. quarterly visits with STI event | 61 | 82 | 36 | 39

ADVERSE EVENTS:
Time Frame: Duration of participants participation, up to 1 year.
Description: The following AEs were recorded at each study visit:
  * All grade 2 and higher hematologic and hepatic laboratory abnormalities that are attributed to doxycycline in the opinion of the site investigator
  * All AEs meeting SAE definition
  * All grade 3 and 4 adverse events judged to be associated with doxycycline (possibly, probably, or definitely related)
  * NOTE: Non-serious adverse events were not collected or reported in participants assigned to a control arm, per protocol.
Groups:
- PrEP Cohort: Doxy PEP: Doxycycline 200mg in addition to standard of care STI testing and treatment - HIV-negative participants on PrEP at time of enrollment or starting PrEP within 30 days of enrollment.
  Doxycycline Hyclate Delayed-Release 200 mg: 200 mg of doxycycline taken by mouth after condomless sexual contact as post exposure prophylaxis (PEP).
  The number of participants assessed for serious and non-serious adverse events excludes those who did not attend any follow-up visits after baseline.
- PrEP Cohort: Control; PLWH: Control: The control arm will consist of standard of care STI testing and treatment - HIV-negative participants on PrEP at time of enrollment or starting PrEP within 30 days of enrollment.
  The number of participants assessed for serious adverse events excludes those who did not attend any follow-up visits after baseline.
- PLWH Cohort: Doxy PEP: Doxycycline 200mg in addition to standard of care STI testing and treatment - People living with HIV Doxycycline Hyclate Delayed-Release 200 mg: 200 mg of doxycycline taken by mouth after condomless sexual contact as post exposure prophylaxis (PEP).
  The number of participants assessed for serious and non-serious adverse events excludes those who did not attend any follow-up visits after baseline.
Arm/Group | PrEP Cohort: Doxy PEP | PrEP Cohort: Control | PLWH Cohort: Doxy PEP | PLWH: Control
All-Cause Mortality (participants affected / at risk) | 0/217 | 0/100 | 0/109 | 0/47
Serious Adverse Events (participants affected / at risk) | 1/217 | 1/100 | 2/109 | 0/47
Other Adverse Events (participants affected / at risk) | 6/217 | 0/0 | 0/109 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PrEP Cohort: Doxy PEP (N=217) | PrEP Cohort: Control (N=100) | PLWH Cohort: Doxy PEP (N=109) | PLWH: Control (N=47)
Cat bite (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Required hospitalization
Testicular torsion (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Required surgery
Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Due to substance use, required hospitalization
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Required hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PrEP Cohort: Doxy PEP (N=217) | PrEP Cohort: Control (N=0) | PLWH Cohort: Doxy PEP (N=109) | PLWH: Control (N=0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) — Grade 3
Elevated ALT (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Grade 2
Headache/migraine (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) — Grade 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-05-27): https://cdn.clinicaltrials.gov/large-docs/23/NCT03980223/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/23/NCT03980223/SAP_001.pdf
  • Informed Consent Form (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/23/NCT03980223/ICF_002.pdf